CLINICAL TRIAL: NCT00168688
Title: The Effects of Prenatal Multi-micronutrient Supplements on Pregnancy Outcome, Peri- and Neonatal Mortality on Maternal and Infant Nutritional Status: A Randomised, Controlled Trial Among Women in Guinea-Bissau
Brief Title: Prenatal Multi-micronutrient Supplementation and Pregnancy Outcome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Royal Veterinary and Agricultural University, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RUF-2001-91057-PREGNUT
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Pregnancy; Birth Weight
Keywords: micronutrient supplementation; pregnancy; birth weight; perinatal mortality
MeSH Terms: conditions — Birth Weight; Perinatal Death

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- FeFol (Active Comparator): Iron (60 mg) and folic acid (400 ug), standard of care
  Interventions: Dietary Supplement: multi micronutrient supplement
- MN1 (Experimental): 1 RDA of 15 micronutrients, including iron (30 mg) and folic acid (400 ug)
  Vitamin A 800 μg RE, Vitamin D 200 IU, Vitamin E 10 mg, Vitamin B1 1.4 mg, Vitamin B2 1.4 mg, Niacin 18 mg, Folic acid 400 μg, Vitamin B6 1.9 mg, Vitamin B12 2.6 μg, Vitamin C 70 mg, Zinc 15 mg, Iron 30 mg, Copper 2.0 mg, Selenium 65 μg, Iodine 150 μg
  Interventions: Dietary Supplement: MN1
- MN2 (Experimental): 2 RDA of 14 micronutrients including iron (30 mg) and folic acid (800 ug)
  Vitamin A 1600 μg RE, Vitamin D 400 IU, Vitamin E 20 mg, Vitamin B1 2.8 mg, Vitamin B2 2.8 mg, Niacin 36 mg, Folic acid 800 μg, Vitamin B6 3.8 mg, Vitamin B12 5.2 μg, Vitamin C 140 mg, Zinc 30 mg, Iron 30 mg, Copper 4.0 mg, Selenium 130 μg, Iodine 300 μg
  Interventions: Dietary Supplement: MN2

INTERVENTIONS:
Dietary Supplement: multi micronutrient supplement
  Arms: FeFol
Dietary Supplement: MN1 — Vitamin A 800 μg RE, Vitamin D 200 IU, Vitamin E 10 mg, Vitamin B1 1.4 mg, Vitamin B2 1.4 mg, Niacin 18 mg, Folic acid 400 μg, Vitamin B6 1.9 mg, Vitamin B12 2.6 μg, Vitamin C 70 mg, Zinc 15 mg, Iron 30 mg, Copper 2.0 mg, Selenium 65 μg, Iodine 150 μg
  Arms: MN1
Dietary Supplement: MN2 — Vitamin A 1600 μg RE, Vitamin D 400 IU, Vitamin E 20 mg, Vitamin B1 2.8 mg, Vitamin B2 2.8 mg, Niacin 36 mg, Folic acid 800 μg, Vitamin B6 3.8 mg, Vitamin B12 5.2 μg, Vitamin C 140 mg, Zinc 30 mg, Iron 30 mg, Copper 4.0 mg, Selenium 130 μg, Iodine 300 μg
  Arms: MN2

SUMMARY:
Prenatal maternal micronutrient supplementation has been suggested as a means to reduce the proportion of low birth weight babies in low-income countries. The effects of prenatal multi-micronutrient supplements on birth weight and perinatal mortality were studied in a randomised controlled trial among 2100 pregnant women in Guinea-Bissau. Women up to 37 weeks pregnant were individually randomised to daily supplements until delivery of A) Iron + folic acid or multi-micronutrients in B) One or C) Two recommended dietary allowances. Secondary outcomes were infant growth and maternal haemoglobin eight weeks after delivery.

DETAILED DESCRIPTION:
Prenatal maternal micronutrient supplementation has been suggested as a means to reduce the proportion of low birth weight babies in low-income countries. The effects of prenatal multi-micronutrient supplements on birth weight and perinatal mortality were studied in a randomised controlled trial among 2100 pregnant women in Guinea-Bissau. Women up to 37 weeks pregnant were individually randomised to daily supplements until delivery of identically looking tablets containing 1) Iron (60 mg) + folate (400 µg), 2) One recommended dietary allowance (RDA) of 5 minerals and 10 vitamins, including iron (30 mg) and folate (400 µg), or 3) Two RDA's of 5 minerals and 10 vitamins, including iron (30 mg) and folate (800 µg). Supplements were provided in known excess at fortnightly home visits until delivery. Compliance was assessed by tablet count.

Women were interviewed about age, civil status, obstetric history and socio-economic status at enrolment. Maternal anthropometry was measured at enrolment, at delivery, and eight weeks after delivery. Maternal malaria parasitaemia and haemoglobin were measured at enrolment and eight weeks after delivery. Maternal status of a wide range of micronutrients was assessed at enrolment and eight weeks after delivery in a sub-cohort of 600 women. Further, survival of the infants will be followed until 3 years of age, within the routines of the Bandim Health Project surveillance system.

Women were provided impregnated bed nets and weekly malaria prophylaxis until delivery. Women with high malaria parasitaemia at enrolment were in addition given a full treatment at enrolment.

Sample size considerations: A sample size of 638 women in each treatment group will be required to detect a reduction in perinatal mortality from 9% to 5% or less in a treatment group using 80% power and a 5% significance level. With an expected loss to follow up of 10%, 2100 women are required. With a sample size of 2100 the study will be able to detect at least 75 g difference, i.e. a 2.5% change in birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

Exclusion Criteria:

* >37 weeks of gestational at enrollment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2100 (Actual)
Dates: Start 2001-01; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Birth weight (<3 days)
Perinatal mortality

SECONDARY OUTCOMES:
Maternal haemoglobin (8 weeks pp)
Maternal anthropometry (8 weeks pp)
Infant growth (8 weeks pp)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Dr. Med, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

REFERENCES:
- [Result] Kaestel P, Michaelsen KF, Aaby P, Friis H. Effects of prenatal multimicronutrient supplements on birth weight and perinatal mortality: a randomised, controlled trial in Guinea-Bissau. Eur J Clin Nutr. 2005 Sep;59(9):1081-9. doi: 10.1038/sj.ejcn.1602215. PMID 16015266